CLINICAL TRIAL: NCT02471924
Title: Predicting Hypotension Related to Spinal Anesthesia for Caesarean Section With Ultrasonography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2015-13
Record Dates: First submitted 2015-06-02; First posted 2015-06-15 (Estimated); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Pregnancy
Keywords: Pregnant women

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Trans thoraciq cardiac ultrasonography (Other): Trans thoraciq cardiac ultrasonography wil be perforfomed for pregnant women having a spinal or spinal-epidural anesthesia for elective caesarean section. All patients are more 18 years old and more 37 weeks pregnancy
  Interventions: Other: Trans thoraciq cardiac ultrasonography

INTERVENTIONS:
Other: Trans thoraciq cardiac ultrasonography — Establish a diagnosis power of the ΔITVAo ( aortic velocity peak )measured with cardiac Trans thoraciq ultrasonography after passiv leg rising to predict hypotension after spinal anesthesia for elective caesarean. Every patients participate for 30 minutes (time to perform the echography). Outside echographic evaluation, medical taking of participating patients will be exactly the same than what is done for all elective caesarean section.

SUMMARY:
Spinal anesthesia is the main technique for caesarean section. This anesthesia is followed by a hypotension in 40% to 90% despite preventing tools. Hypotension is responsible of foetale and maternal suffering. It would be interesting to have a tool that could detect patient who are at risk to have hypotension.This study consist in measuring variations of under aortic velocity peak (ΔITVAo) which estimate the modification of the cardiac output by Trans thoraciq echography.

DETAILED DESCRIPTION:
Spinal anesthesia is the main technique for caesarean section. This anesthesia is followed by a hypotension in 40% to 90% despite preventing tools (fluid challenge and vasoactives drugs). Hypotension is responsible of foetale and maternal suffering. Fluid challenge is able to upgrade cardiac output for some patient, for some other it is unusefull or it can deteriorate it. Actually fluid challenge is not individualized. It would be interesting to have a tool that could detect patient who are at risk to have hypotension.

Trans thoraciq echography is an easy non invading tool. Dynamic criteria which is recognized for predicting vascular filling , with spontaneus breathing, is the passive leg rising (PLR). PLR mime à vascular filling of 500 ml. Modification of this cardiac outpout is measured whith the echocardiograph. This consist in measuring variations of under aortic velocity peak (ΔITVAo) which estimate the modification of the cardiac output.

ELIGIBILITY:
Inclusion Criteria:

* Included patient are all women having a spinal or spinal-epidural anesthesia for elective caesarean section. All patients are more 18 years old and more 37 weeks pregnancy.

Physical statut score (ASA):1 or 2

Exclusion Criteria:

* Woman presenting a contraindication to the spinal epidural anesthesia : constitutional or acquired disorder of the haemostasis
* allergy in the local anesthetics,
* infectious context (hypertherm > 38.5 ° C)

  · cardiac, right or left Insufficiency
* eclamptic toxemia

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-06-17 (Actual); Primary Completion 2017-02-20 (Actual); Study Completion 2017-10-10 (Actual)

PRIMARY OUTCOMES:
Establish a diagnosis power of the ΔITVAo measured with cardiac ultrasonography after passiv leg rising to predict hypotension after spinal anesthesia for elective caesarean. | 1 year
  ITVAo corresponds to the variation of complete time speed under aortic between the measure position half seat and the measure of the ITVAo during the test of rise of passive leg.
  ITVAo is a reflection of the variation of the volume of systolic ejection. The variation of the volume of systolic ejection led during the test of rise of passive leg, measured in cardiac ultrasound , predicts the answer to the vascular filling at patients of resuscitation
  The definition retained for the low blood pressure is a fall of 20 % of the mean arterial blood pressure of base in the first 15 minutes which follow the spinal anesthesia. The basic value of the mean arterial blood pressure is defined as the average of 3 mean arterial blood pressure measures in 3 minutes apart in dorsal decubitus before the practice of the spinal anesthesia

SECONDARY OUTCOMES:
Estimate if ΔITVAo is linked to an increase in vasoactiv drugs | 1 year
Estimate if ΔITVAo is linked to fœtal suffering (low acido basic statues in blood section and low APGAR score) | 1 year
Estimate if other echographic measures are linked to hypotension after spinal anesthesia | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Carole BECHIS, MD, Principal Investigator — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] Zieleskiewicz L, Noel A, Duclos G, Haddam M, Delmas A, Bechis C, Loundou A, Blanc J, Mignon A, Bouvet L, Einav S, Bourgoin A, Leone M. Can point-of-care ultrasound predict spinal hypotension during caesarean section? A prospective observational study. Anaesthesia. 2018 Jan;73(1):15-22. doi: 10.1111/anae.14063. Epub 2017 Oct 7. PMID 28986931